CLINICAL TRIAL: NCT03339089
Title: Real-world Effectiveness of Adalimumab on Health Outcomes in Chinese Patients With Immune-Mediated Inflammatory Diseases
Acronym: ADMIT
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-828
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Ankylosing Spondylitis (AS); Psoriasis; Rheumatoid Arthritis (RA)
Keywords: rheumatoid arthritis; plaque psoriasis; ankylosing spondylitis; Immune-Mediated Inflammatory Diseases; Chinese Patients
MeSH Terms: conditions — Spondylitis, Ankylosing; Psoriasis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Participants with Rheumatoid Arthritis (RA): This group/ cohort includes participants with RA.
- Participants with Plaque Psoriasis (Ps): This group/ cohort includes participants with Ps.
- Participants with Ankylosing spondylitis (AS): This group/ cohort includes participants with AS.

SUMMARY:
The objective of this study is to evaluate the effect of adalimumab on health outcomes in participants with rheumatoid arthritis, ankylosing spondylitis and plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of rheumatoid arthritis, ankylosing spondylitis or plaque psoriasis
* Decision to initiate Humira® treatment in accordance with routine medical practice and in compliance with eligibility for adalimumab based on the local label
* Prior to any study-specific procedures, participant has voluntarily signed the authorization (or informed consent where applicable) to disclose and use anonymized personal health information after participate in this research.

Exclusion Criteria:

* Inadequate response to previous standard treatment with anti-tumor necrosis factor (TNF) biological agent according to the physician's clinical judgment.
* Participant has been treated with adalimumab within 70 days (five half-lives) prior to the Baseline Visit.
* Participants discontinued due to adverse drug reaction of previous adalimumab treatment.
* Participants who fulfill any of the contraindications as per adalimumab label in China.
* Participants, who in the clinician's view, may not be able to comply with the study requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese participants diagnosed with rheumatoid arthritis, ankylosing spondylitis or plaque psoriasis, for whom adalimumab (Humira®) treatment has already been decided as per local label, will be recruited from within the clinical setting of each rheumatologist or dermatologist participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in EuroQoL-5 Dimension (EQ-5D) index score up to Week 24 | From Week 0 to Week 24
  The European quality of life-5 dimensions (EQ-5D) is a simple, easy to administer, standardized and self-report instrument for health status, which is applicable to a wide range of health conditions and treatment.

SECONDARY OUTCOMES:
Assessing drug persistence | Up to Week 52
  This is measured using drug survival rate.
Change from baseline in Healthcare Resource Utilization (HCRU) | From Week 0 to Week 52
  This is assessed using the HCRU questionnaire.
Change from baseline in Work productivity and Activity Impairment questionnaire - Specific Health Problem (WPAI-SHP) in participants with Ankylosing spondylitis (AS) | Up to Week 52
  WPAI questionnaire will be used to measure work absenteeism, work presenteeism, and daily activity impairment.
Change from Baseline in Dermatology Life Quality Index (DLQI) in participants with Psoriasis (Ps) | Up to Week 52
  The Dermatology Life Quality Index (DLQI) is the most commonly used quality of life (QoL) assessment tool in psoriasis clinical research.
Change from baseline in Work productivity and Activity Impairment questionnaire - Specific Health Problem (WPAI-SHP) in participants with Rheumatoid Arthritis (RA) | Up to Week 52
  WPAI questionnaire will be used to measure work absenteeism, work presenteeism, and daily activity impairment.
Change from baseline in Clinical Disease Activity Index (CDAI) in participants with Rheumatoid Arthritis (RA) | Up to Week 52
  The CDAI is used to evaluate disease activity.
Percentage of participants achieving low disease activity (CDAI 2.8-10) in participants with Rheumatoid Arthritis (RA) | Up to Week 52
  The CDAI is used to evaluate disease activity.
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in participants with Ankylosing spondylitis (AS) | Up to Week 52
  BASDAI score is determined using a simple, self-reported questionnaire.
Percentage of participants achieving remission (CDAI<=2.8) in participants with Rheumatoid Arthritis (RA) | Up to Week 52
  The CDAI is used to evaluate disease activity.
Change from baseline in EQ-5D Visual analog scale (VAS) | From Week 0 to Week 52
  It is a patient-reported outcome (PRO) questionnaires used to assess quality of life (QoL).
Change from baseline in EQ-5D index score up to Week 52 | From Week 0 to Week 52
  The European quality of life-5 dimensions (EQ-5D) is a simple, easy to administer, standardized and self-report instrument for health status, which is applicable to a wide range of health conditions and treatment.
Proportion of participants achieving Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 response in participants with Ankylosing spondylitis (AS) | Up to Week 52
  BASDAI score is determined using a simple, self-reported questionnaire.
Change from baseline in Psoriasis Area and Severity Index (PASI) in participants with Psoriasis (Ps) | Up to Week 52
  PASI provides a quantitative assessment of psoriasis disease state.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- China (10):
  - Shenzhen Futian Hospital for rheumatic Diseases /ID# 209340, Shenzhen, Guangdong
  - AbbVie China /ID# 164373, Shanghai, Shanghai Municipality
  - The First affiliated hospital of chengdu medical university /ID# 210745, Chengdu, Sichuan
  - Zhejiang Province People's Hospital /ID# 209342, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital /ID# 210820, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing /ID# 213686, Jiaxing, Zhejiang
  - The Second Hospital of Jiaxing /ID# 210744, Jiaxing, Zhejiang
  - Jinhua Municipal Central Hospital /ID# 209339, Jinhua, Zhejiang
  - Sichuan Provincial orthopedic hospital /ID# 209341, Chengdu
  - West China Hospital, SCU West China School of Medicine, SCU /ID# 209333, Chengdu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P16-828&Latitude=&Longitude=&LocationName=#additional-resources-section